CLINICAL TRIAL: NCT05045716
Title: An Open-label, Parallel-group, Randomized Study to Evaluate the Absolute Bioavailability of Single Dose Subcutaneous Administration of Lecanemab in Healthy Subjects
Brief Title: A Study of Subcutaneous Lecanemab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BAN2401-A001-004
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers
Keywords: Lecanemab; Bioavailability; Subcutaneous
MeSH Terms: interventions — lecanemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lecanemab 10 mg/kg (Experimental): Participants will receive lecanemab 10 milligram per kilogram (mg/kg), as single dose IV infusion over approximately 1 hour on Day 1.
  Interventions: Drug: Lecanemab
- Lecanemab 700 mg (Experimental): Participants will receive lecanemab 700 milligram (mg), as single fixed dose SC injection in the abdomen on Day 1.
  Interventions: Drug: Lecanemab

INTERVENTIONS:
Drug: Lecanemab — Lecanemab IV infusion.
  Other Names: BAN2401
  Arms: Lecanemab 10 mg/kg
Drug: Lecanemab — Lecanemab SC injection.
  Other Names: BAN2401
  Arms: Lecanemab 700 mg

SUMMARY:
The primary purpose of this study is to determine the absolute bioavailability and pharmacokinetic (PK) profile of a single dose of lecanemab when administered subcutaneously (SC) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

1. Non-smoking, male or female, age greater than or equal to (>=) 18 years and less than or equal to (<=) 65 years old at the time of informed consent. To be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing.
2. Japanese participants (age >=20 years) must have been born in Japan of Japanese parents and Japanese grandparents, must have lived no more than 5 years outside of Japan, and must not have changed their lifestyle or habits, including diet, while living outside of Japan.
3. Body Mass Index (BMI) >=18 and less than (<) 30 kilogram per square meter (kg/m^2) at screening.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing.
2. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism
3. Exposure within the last 14 days before dosing to an individual with confirmed or probable corona virus disease-2019 (COVID-19) or symptoms within the last 14 days that are on the most recent Centers for Disease Control and Prevention list of COVID symptoms or any other reason to consider the participant at potential risk for COVID-19 infection
4. Participants who had received COVID vaccine but are not 14 days post full vaccination before dosing
5. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5 half-lives of the other investigational drug, whichever is longer, preceding informed consent
6. Prior exposure to lecanemab
7. Hypersensitivity to lecanemab or any of the excipients, or to any monoclonal antibody treatment

NOTE-Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
AUC(0-t): Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration for Lecanemab | Days 0-50
AUC(0-72h): Area Under the Serum Concentration-time Curve From Time Zero to 72 Hours Post End of Intravenous (IV) Infusion or SC Administration for Lecanemab | 0-72 hours
AUC(0-inf): Area Under the Serum Concentration-time Curve From Time Zero to Time Extrapolated to Infinity for Lecanemab | Days 0-50
F: Absolute Bioavailability of SC Formulation for Lecanemab | Days 0-50
  Absolute bioavailability (F) = [AUC(0-inf) SC*Dose (IV)]/[AUC(0-inf) IV*Dose (SC)]. IV dose will be based on total dose (mg) infused.
Cmax: Maximum Observed Serum Concentration for Lecanemab | Days 0-50
Tmax: Time to Reach Maximum Serum Concentration for Lecanemab | Days 0-50
T1/2: Terminal Elimination Half-life for Lecanemab | Days 0-50

SECONDARY OUTCOMES:
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) | Baseline up to Day 50
Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters | Baseline up to Day 22
  Clinical laboratory parameters will include hematology, blood chemistry, and urinalysis.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values | Baseline up to Day 50
  Vital signs parameters will include diastolic and systolic blood pressure (BP), pulse, respiratory rate, body temperature and body weight.
Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings | Baseline up to Day 50
Number of Participants With Positive and Negative Anti-drug Antibody (ADA) for Lecanemab | Baseline Up to Day 50
  ADA will be measured using validated electrochemiluminescent immunoassay (ECL) methods.
Number of Participants With Neutralizing Antibodies (NAb) for Lecanemab | Baseline up to Day 50
  NAb will be measured using validated ECL methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.